CLINICAL TRIAL: NCT03042468
Title: Phase I/ll Dose-escalation Study of Fractionated Dose 177Lu-PSMA-617 for Progressive Metastatic Castration Resistant Prostate Cancer
Brief Title: Phase I Dose-escalation Study of Fractionated 177Lu-PSMA-617 for Progressive Metastatic CRPC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1609017542; PSMA-617 (Other: Weill Cornell Medical College)
Record Dates: First submitted 2017-01-19; First posted 2017-02-03 (Estimated); Results first posted 2022-12-13 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto; gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): 1. 177Lu-PSMA-617 [50mCi (1.85GBq) - 300mCi (11.1GBq)] intravenous X2 doses, 2 weeks apart (Visit 1 and 2)
  2. 68Ga-PSMA-HBED-CC [5 ±2mCi or 185 ±74MBq] intravenous during screening and at 12 weeks with standard imaging
  Interventions: Drug: 177Lu-PSMA-617; Drug: 68Ga-PSMA-HBED-CC

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — 177Lu-PSMA-617 [50mCi (1.85GBq) - 300mCi (11.1GBq)] intravenous X2 doses, 2 weeks apart (Visit 1 and 2)
Drug: 68Ga-PSMA-HBED-CC — 68Ga-PSMA-HBED-CC [5 ±2mCi or 185 ±74MBq] intravenous during screening and at 12 weeks with standard imaging

SUMMARY:
The purpose of this study is to find the highest dose level of the study drug, 177Lu-PSMA-617 that can be given without severe side effects for advanced prostate cancer.

DETAILED DESCRIPTION:
Phase I dose escalation study with 177Lu-PSMA-617 using dose fractionation regimen will be performed in patients with documented progressive metastatic CRPC. The cumulative 177Lu dose [100 mCi (3.7 GBq) - 600 mCi (22.2 GBq)] will be escalated in up to 6 different dose levels (3 + 3 study design). Additional 10 subjects will be enrolled at the MTD dose level to further assess safety and tolerability and to obtain a preliminary assessment of efficacy. The study will enroll adult males 18 years of age or older with documented progressive metastatic CRPC. The primary objectives are: - To determine the dose limiting toxicity (DLT) of fractionated dose of 177Lu-PSMA-617 - To determine the maximal tolerated and recommended phase II dose of 177Lu-PSMA-617 in a 2-week dose-fractionation regimen Subjects will receive the following study interventions:

1. 177Lu-PSMA-617 [50mCi (1.85GBq) - 300mCi (11.1GBq)] intravenous X2 doses, 2 weeks apart (Visit 1 and 2)
2. 68Ga-PSMA-HBED-CC [5 ±2mCi or 185 ±74MBq] intravenous during screening and at 12 weeks with standard imaging Subjects will be on this study from screening to end of study (day 85).

The treatment phase comprises of 8 visits over 12 weeks. Patients will be followed until death for survival assessment. Patients removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event. All tests and procedures performed on this study are routine and standard of care except: 68Ga-PSMA-HBED-CC PET/CT scan, administration of investigational agent 177Lu-PSMA-617, research blood samples (CTCs for research, cell-free DNA sample), and PSMA testing on archive tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of prostate
2. Documented progressive metastatic CRPC based on Prostate Cancer Working Group 3 (PCWG3) criteria, which includes at least one of the following criteria:

   * PSA progression
   * Objective radiographic progression in soft tissue
   * New bone lesions
3. ECOG performance status of 0-2
4. Have serum testosterone < 50 ng/dL. Subjects must continue primary androgen deprivation with an LHRH/GnRH analogue (agonist/antagonist) if they have not undergone orchiectomy.
5. Have previously been treated with at least one of the following:

   * Androgen receptor signaling inhibitor (such as enzalutamide)
   * CYP 17 inhibitor (such as abiraterone acetate)
6. Have previously received taxane chemotherapy, been determined to be ineligible for taxane chemotherapy by their physician, or refused taxane chemotherapy.
7. Age > 18 years
8. Patients must have normal organ and marrow function as defined below:

   * Absolute neutrophil count >2,000 cells/mm3
   * Hemoglobin ≥9 g/dL (independent of transfusion and/or growth factors within 1 month prior to registration)
   * Platelet count >150,000 x 109/uL (independent of transfusion and/or growth factors within 3 months prior to randomization)
   * Serum creatinine <1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min/1.73 m2 by Cockcroft-Gault
   * Serum total bilirubin <1.5 x ULN (unless due to Gilbert's syndrome in which case direct bilirubin must be normal
   * Serum AST and ALT <1.5 x ULN
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Use of investigational drugs or implantation of investigational medical device ≤4 weeks of Cycle 1, Day 1 or current enrollment in investigational drug or device study
2. Prior systemic beta-emitting bone-seeking radioisotopes
3. Brain metastases or leptomeningeal disease
4. History of deep vein thrombosis and/or pulmonary embolus within 1 month of study entry
5. Other serious illness(es) involving the cardiac, respiratory, CNS, renal, hepatic or hematological organ systems which might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study
6. Radiation therapy for treatment of PCa ≤4 weeks of Day 1 Cycle 1
7. Patients on stable dose of bisphosphonates or denosumab, which have been started no less than 4 weeks prior to treatment start, may continue on this medication, however patients are not allowed to initiate bisphosphonate/Denosumab therapy during the DLT-assessment period of the study.
8. Having partners of childbearing potential and not willing to use a method of birth control deemed acceptable by the principle investigator and chairperson during the study and for 1 month after last study drug administration
9. Currently active other malignancy other than non-melanoma skin cancer. Patients are considered not to have "currently active" malignancy if they have completed any necessary therapy and are considered by their physician to be at less than 30% risk of relapse.
10. Known history of known myelodysplastic syndrome

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12; Primary Completion 2021-09-30 (Actual); Study Completion 2026-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Tagawa, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Tulane Cancer Center Clinic, New Orleans, Louisiana
  - Weill Cornell Medical College, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vlachostergios PJ, Niaz MJ, Skafida M, Mosallaie SA, Thomas C, Christos PJ, Osborne JR, Molina AM, Nanus DM, Bander NH, Tagawa ST. Imaging expression of prostate-specific membrane antigen and response to PSMA-targeted beta-emitting radionuclide therapies in metastatic castration-resistant prostate cancer. Prostate. 2021 Apr;81(5):279-285. doi: 10.1002/pros.24104. Epub 2021 Jan 19. PMID 33465252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at at Weill Cornell Medicine New York Presbyterian and Tulane Medical Center.
Groups:
- 177Lu-PSMA-617 Cohort 1: Cohort 1: Participants were administered of 177Lu-PSMA-617 once at the dose level of 50mCi (1.85GBq) via intravenous infusion (IV) in two doses two weeks apart at Visits 1 and 2. Participants were then followed until death for survival assessment
- 177Lu-PSMA-617 Cohort 2: Cohort 2: Participants were administered of 177Lu-PSMA-617 once at the dose level of 100mCi (3.7GBq) via intravenous infusion (IV) in two doses two weeks apart at Visits 1 and 2. Participants were then followed until death for survival assessment
- 177Lu-PSMA-617 Cohort 3: Cohort 3: Participants were administered of 177Lu-PSMA-617 once at the dose level of 200mCi (7.4GBq) via intravenous infusion (IV) in two doses two weeks apart at Visits 1 and 2. Participants were then followed until death for survival assessment
- 177Lu-PSMA-617 Cohort 4: Cohort 4: Participants were administered of 177Lu-PSMA-617 once at the dose level of 250mCi (9.25GBq) via intravenous infusion (IV) in two doses two weeks apart at Visits 1 and 2. Participants were then followed until death for survival assessment
- 177Lu-PSMA-617 Cohort 5: Cohort 5: Participants were administered of 177Lu-PSMA-617 once at the dose level of 300mCi (11.1GBq) via intravenous infusion (IV) in two doses two weeks apart at Visits 1 and 2. Participants were then followed until death for survival assessment
- Dose Expansion Cohort: Participants followed Cohort 5 and were administered 177Lu-PSMA-617 once at the dose level of 300mCi (11.1GBq) via intravenous infusion (IV) in two doses two weeks apart at Visits 1 and 2. Participants were then followed until death for survival assessment.
Period: Overall Study
Arm/Group | 177Lu-PSMA-617 Cohort 1 | 177Lu-PSMA-617 Cohort 2 | 177Lu-PSMA-617 Cohort 3 | 177Lu-PSMA-617 Cohort 4 | 177Lu-PSMA-617 Cohort 5 | Dose Expansion Cohort
Started | 6 | 6 | 5 | 6 | 6 | 21
Completed | 6 | 5 | 4 | 6 | 5 | 19
Not Completed | 0 | 1 | 1 | 0 | 1 | 2
Not completed — Death | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 177Lu-PSMA-617 Cohort 1 | 177Lu-PSMA-617 Cohort 2 | 177Lu-PSMA-617 Cohort 3 | 177Lu-PSMA-617 Cohort 4 | 177Lu-PSMA-617 Cohort 5 | Dose Expansion Cohort | Total
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 21 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 2 | 0 | 3 | 4 | 10
  >=65 years | 6 | 5 | 3 | 6 | 3 | 17 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 5 | 6 | 6 | 21 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 0 | 0 | 2 | 4
  White | 4 | 4 | 4 | 6 | 6 | 19 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose Limiting Toxicity (DLT) of Fractionated Dose of 177Lu-PSMA-617
Description: Proportion of subjects experiencing a dose limiting toxicity (DLT) of fractionated dose of 177Lu-PSMA-617 by using 3+3 dose escalation was assessed.
Time Frame: Assessed throughout the DLT period, up to 92 days after starting study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 177Lu-PSMA-617 Cohort 1 | 177Lu-PSMA-617 Cohort 2 | 177Lu-PSMA-617 Cohort 3 | 177Lu-PSMA-617 Cohort 4 | 177Lu-PSMA-617 Cohort 5 | Dose Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 21
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects That Achieved Cumulative Maximum Tolerated Dose (MTD) Phase II Dose of 177Lu-PSMA-617
Description: This outcome is measuring the number of subjects that achieved MTD. MTD is defined as the highest dose level with an observed incidence of DLT in no more than one out of six patients treated at a particular dose level. If no DLTs were experienced, then a recommended phase II dose was determined in 2-wk dose-fractionation regimen by using a 3+3 dose escalation design, as no MTD was observed.
Time Frame: from first dose of study drug to at least 12 weeks of subsequent follow-up evaluations, up to 92 days
Measure: Count of Participants; unit: Participants
Arm/Group | 177Lu-PSMA-617 Cohort 1 | 177Lu-PSMA-617 Cohort 2 | 177Lu-PSMA-617 Cohort 3 | 177Lu-PSMA-617 Cohort 4 | 177Lu-PSMA-617 Cohort 5 | Dose Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 21
Participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Recommended Phase II Dose of 177Lu-PSMA-617 in a 2-week Dose-fractionation Regimen
Description: Recommended Phase II dose was determined based on the results of the Phase I portion of the study. Since no Maximum Tolerated Dose was achieved given that no Dose Limiting Toxicities occurred, the Recommended Phase II dose was determined based on the Cohort 5 dose.
Time Frame: Duration of Phase I, up to 47 months
Measure: Number; unit: mci
Groups:
- All Phase 1 Subjects: 1. 177Lu-PSMA-617 [50mCi (1.85GBq) - 300mCi (11.1GBq)] intravenous X2 doses, 2 weeks apart (Visit 1 and 2)
  2. 68Ga-PSMA-HBED-CC [5 ±2mCi or 185 ±74MBq] intravenous during screening and at 12 weeks with standard imaging
  177Lu-PSMA-617: 177Lu-PSMA-617 [50mCi (1.85GBq) - 300mCi (11.1GBq)] intravenous X2 doses, 2 weeks apart (Visit 1 and 2)
  68Ga-PSMA-HBED-CC: 68Ga-PSMA-HBED-CC [5 ±2mCi or 185 ±74MBq] intravenous during screening and at 12 weeks with standard imaging
Arm/Group | All Phase 1 Subjects
Number analyzed (Participants) | 29
mci | 300

4. Secondary Outcome: The Rate of PSA Decline Following Fractionated 177Lu-PSMA-617
Description: Proportion of patients with PSA decline following treatment (fractionated 177Lu-PSMA-617) with the RP2D of fractionated dose 177Lu-PSMA-617 (Phase II). PSA response will be determined by comparing the PSA levels after therapy to the baseline, pre-treatment PSA.
Time Frame: from baseline visit to short term follow up visit, approximately 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 177Lu-PSMA-617 Cohort 1 | 177Lu-PSMA-617 Cohort 2 | 177Lu-PSMA-617 Cohort 3 | 177Lu-PSMA-617 Cohort 4 | 177Lu-PSMA-617 Cohort 5 | Dose Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 21
Participants | 5 | 3 | 3 | 6 | 6 | 21

5. Secondary Outcome: Count of Patients That Had a Radiographic Response Rate Measured by RECIST 1.1 With PCWG3 Modifications
Time Frame: From start of study to progression of disease with at least 12 weeks of subsequent follow-up evaluations, up to 54 months
Population: Only evaluable subjects were analyzed for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | 177Lu-PSMA-617 Cohort 1 | 177Lu-PSMA-617 Cohort 2 | 177Lu-PSMA-617 Cohort 3 | 177Lu-PSMA-617 Cohort 4 | 177Lu-PSMA-617 Cohort 5 | Dose Expansion Cohort
Number analyzed (Participants) | 6 | 0 | 1 | 1 | 4 | 5
Participants | 4 | 0 | 1 | 1 | 1 | 3

6. Secondary Outcome: Progression-free Survival Measured by PCWG3 (Prostate Cancer Working Group3) Criteria
Description: Progression Free Survival, with progression determined based by Radiographic and Biochemical response. Biochemical response was assessed by comparing the PSA levels after therapy to the baseline, pre-treatment PSA. Declines of ≥ 30% confirmed by a second PSA value ≥2 weeks later, are reported.
Time Frame: Duration of time on study, from baseline to last follow up visit, up to 54 months
Measure: Mean (Full Range); unit: days
Arm/Group | 177Lu-PSMA-617 Cohort 1 | 177Lu-PSMA-617 Cohort 2 | 177Lu-PSMA-617 Cohort 3 | 177Lu-PSMA-617 Cohort 4 | 177Lu-PSMA-617 Cohort 5 | Dose Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 21
days | 95 [42 to 118] | 147 [14 to 429] | 119 [14 to 357] | 188 [83 to 449] | 99 [13 to 265] | 176 [14 to 1145]

7. Secondary Outcome: Number of CTC Count Responders
Description: Changes in CTC count as measured by CellSearch and the rate of favorable CTC count and LDH at 12 weeks following fractionated 177Lu-PSMA-617.
  All subjects in this study will get blood samples drawn (at screening and EOS visit) for CTC enumeration by CellSearch methodology. Participants whose CTC counts drop to less than 5 or stay below 5 (responders) vs. those who remain at least 5 or above (non-responders) at EOS visit are analyzed.
Time Frame: Duration of study, from screening to EOS visit, up to 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- 77Lu-PSMA-617 Cohort 5: Cohort 5: Participants were administered of 177Lu-PSMA-617 once at the dose level of 300mCi (11.1GBq) via intravenous infusion (IV) in two doses two weeks apart at Visits 1 and 2. Participants were then followed until death for survival assessment
Arm/Group | 177Lu-PSMA-617 Cohort 1 | 177Lu-PSMA-617 Cohort 2 | 177Lu-PSMA-617 Cohort 3 | 177Lu-PSMA-617 Cohort 4 | 77Lu-PSMA-617 Cohort 5 | Dose Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 21
Participants | 4 | 4 | 4 | 2 | 4 | 21

8. Secondary Outcome: Overall Survival Following Fractionated 177Lu-PSMA-617
Description: Overall survival was defined as the time from start of 177Lu-PSMA-617 to the date of death from any cause, or last date of follow up.
Time Frame: Up to 5 years
Measure: Mean (Full Range); unit: days
Groups:
- Dose Expasnion Cohort: Participants followed Cohort 5 and were administered 177Lu-PSMA-617 once at the dose level of 300mCi (11.1GBq) via intravenous infusion (IV) in two doses two weeks apart at Visits 1 and 2. Participants were then followed until death for survival assessment.
Arm/Group | 177Lu-PSMA-617 Cohort 1 | 177Lu-PSMA-617 Cohort 2 | 177Lu-PSMA-617 Cohort 3 | 177Lu-PSMA-617 Cohort 4 | 177Lu-PSMA-617 Cohort 5 | Dose Expasnion Cohort
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 21
days | 385 [156 to 554] | 607 [57 to 1471] | 368 [51 to 763] | 743 [248 to 1595] | 409 [84 to 751] | 478 [110 to 1617]

9. Secondary Outcome: Count of Participants That Experience an Adverse Event
Time Frame: From screening to end of study visit, up to 54 months
Measure: Count of Participants; unit: Participants
Arm/Group | 177Lu-PSMA-617 Cohort 1 | 177Lu-PSMA-617 Cohort 2 | 177Lu-PSMA-617 Cohort 3 | 177Lu-PSMA-617 Cohort 4 | 177Lu-PSMA-617 Cohort 5 | Dose Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 21
Participants | 6 | 6 | 5 | 6 | 6 | 21

ADVERSE EVENTS:
Time Frame: Adverse events collected during the duration of the study, from start of study to end of study, up to 5 years.
Description: Patients who passed away during the follow up period were also included.
Arm/Group | 177Lu-PSMA-617 Cohort 1 | 177Lu-PSMA-617 Cohort 2 | 177Lu-PSMA-617 Cohort 3 | 177Lu-PSMA-617 Cohort 4 | 177Lu-PSMA-617 Cohort 5 | Dose Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 6/6 | 6/6 | 5/5 | 5/6 | 6/6 | 19/21
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 2/5 | 1/6 | 0/6 | 3/21
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 5/5 | 6/6 | 6/6 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 177Lu-PSMA-617 Cohort 1 (N=6) | 177Lu-PSMA-617 Cohort 2 (N=6) | 177Lu-PSMA-617 Cohort 3 (N=5) | 177Lu-PSMA-617 Cohort 4 (N=6) | 177Lu-PSMA-617 Cohort 5 (N=6) | Dose Expansion Cohort (N=21)
Bacteremia (Blood and lymphatic system disorders) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower Extremity Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death due to disease progression (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 177Lu-PSMA-617 Cohort 1 (N=6) | 177Lu-PSMA-617 Cohort 2 (N=6) | 177Lu-PSMA-617 Cohort 3 (N=5) | 177Lu-PSMA-617 Cohort 4 (N=6) | 177Lu-PSMA-617 Cohort 5 (N=6) | Dose Expansion Cohort (N=21)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 6 (6) | 6 (6) | 5 (5) | 6 (6) | 6 (6) | 17 (17)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 4 (4) | 3 (3) | 2 (2) | 4 (4)
Xerostemia (General disorders) | 3 (3) | 5 (5) | 2 (2) | 6 (6) | 6 (6) | 14 (14)
Pain (General disorders) | 6 (6) | 6 (6) | 5 (5) | 5 (5) | 6 (6) | 19 (19)
Fatigue (General disorders) | 6 (6) | 6 (6) | 5 (5) | 6 (6) | 6 (6) | 19 (19)
Nausea (General disorders) | 3 (3) | 0 (0) | 3 (3) | 4 (4) | 2 (2) | 14 (14)
AST increased (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 5 (5)
High Creatinine (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 7 (7)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALP increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALT increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 5 (5) | 3 (3) | 1 (1) | 5 (5)
Arthralgias (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bells palsy (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cough (General disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Death due to progression (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysguesia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0
Facial trauma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypocalcemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle weakness LL (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Nocturia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritendinitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (white blood cell count decreased) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT03042468/Prot_SAP_000.pdf